CLINICAL TRIAL: NCT06243991
Title: The Effect Of High And Low Molecular Weight Sodium Hyaluronic Acid Eye Drops On Corneal Recovery After Crosslinking
Brief Title: The Effect Of High And Low Molecular Weight Sodium Hyaluronic Acid Eye Drops After Crosslinking
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.86
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Keratoconus
Keywords: Corneal crosslinking, corneal nerve regeneration, in-vivo corneal confocal microscopy, sodium hyaluronic acid,; high molecular weight hyaluronic acid
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Nineteen patiens (20 eyes) received topical polyvinyl alcohol (Refresh, Allergan, Dublin, Ireland) three times daily until epithelial defect closure after CXL in control group.
  Interventions: Device: in vivo Corneal Confocal Microscopy; Diagnostic Test: Corneal Sensitivity; Device: Non invasive tear break up time; Diagnostic Test: Ocular Surface Disease Index Qestionnaire; Device: Corneal tomography
- LMW-HA group: Twenty-two patiens (23 eyes) received topical LMW-HA (Thealose Duo®, Thea, Clermont-Ferrand, France) three times daily for 12 months.
  Interventions: Device: in vivo Corneal Confocal Microscopy; Diagnostic Test: Corneal Sensitivity; Device: Non invasive tear break up time; Diagnostic Test: Ocular Surface Disease Index Qestionnaire; Device: Corneal tomography
- HMW-HA group: Seventeen patiens (20 eyes) received topical HMW-HA (Comfort Shield®, i.com medical GmbH, Munich, Germany) three times daily for 12 months.
  Interventions: Device: in vivo Corneal Confocal Microscopy; Diagnostic Test: Corneal Sensitivity; Device: Non invasive tear break up time; Diagnostic Test: Ocular Surface Disease Index Qestionnaire; Device: Corneal tomography

INTERVENTIONS:
Device: in vivo Corneal Confocal Microscopy — CCM was performed using the Heidelberg Retinal Tomograph 3 with the Rostock Cornea Module (HRT3-RCM, Heidelberg Engineering GmbH, Germany) under topical anesthesia. A viscous gel (Viscotears, Novartis Pharmaceuticals UK) served as a coupling agent between the cornea and the applanation cap. The subjects were instructed to focus on the fixation light with the unexamined eye to ensure proper positioning. Five high-quality images of the SNP were selected and analyzed using the automated tracing of nerve fibers program (ACCMetrics, M.A. Dabbah, Imaging Science and Biomedical Engineering, Manchester, England).
Diagnostic Test: Corneal Sensitivity — Corneal sensitivity was evaluated using a Cochet-Bonnet esthesiometer (Luneau Ophtalmologue, Chartres, France), comprising a nylon filament measuring 60 mm in length and 0.12 mm in diameter. Participants were instructed to maintain a forward gaze while the esthesiometer gently made perpendicular contact. The procedure involved gradually decreasing the filament length in 5 mm increments, starting from 60 mm, until the initial response from the subject was detected.
Device: Non invasive tear break up time — Noninvasive tear break-up time (NI-TBUT) was assessed using a Sirius Scheimpflug camera (CSO, Florence, Italy) and the device automatically provided the average NI-TBUT value
Diagnostic Test: Ocular Surface Disease Index Qestionnaire — The Ocular surface disease index (OSDI) questionnaire consists of a total of 12 questions categorized into three subscales as follows: ocular symptoms, vision-related function, and environmental triggers. Each patient is asked to rate the symptoms on a 5-point scale ranging from never (0 score) to always (4 score) for every question in the questionnaire. The fourth and fifth questions in the first section, concerning blurred vision and reduced vision symptoms, were excluded from the questionnaire as these symptoms may already be present in patients with keratoconus disease. The total OSDI score was calculated according to the formula: OSDI = [(sum of scores for all questions answered) × 100] / [(total number of questions answered) × 4].
Device: Corneal tomography — Scheimpflug-tomography device (Pentacam, OCULUS, Wetzlar, Germany) was used for measurement of keratometric values.

SUMMARY:
Purpose: The objective of this investigation was to assess the impact of eye drops containing high molecular weight hyaluronic acid (HMW-HA) and low molecular weight hyaluronic acid (LMW-HA) on corneal nerve regeneration, dendritic cell (DC) density, corneal sensitivity (CS), and ocular surface parameters in patients with keratoconus following corneal crosslinking (CXL).

Methods: Sixty-three eyes of 55 keratoconus patients were randomized to instill eye drops containing HMW-HA (n: 20) for 12 months, LMW-HA (n:23) for 12 months and polyvinyl alcohol (n: 20) until the epithelial defect closure in the control group after CXL. Subbasal nerve plexsus (SNP) was imaged with corneal confocal microscopy (CCM) and ACCMetrics program was used to quantify corneal nerve fiber density (CNFD), corneal nerve fiber length (CNFL), corneal nerve fiber branching density (CNBD) and corneal nerve fiber total branching density (CTBD). DC density was calculated with Image J software. CS was measured using the Cochet-Bonnet esthesiometer. Ocular Surface Disease Index (OSDI) questionnaire, non-invasive break-up time (NI-TBUT) were evaluated. All measurements were performed before CXL and postoperatively after 1, 3, 6 and 12 months.

DETAILED DESCRIPTION:
This study assessed individuals aged 18 and above diagnosed with keratoconus and scheduled for epithelium-off CXL. A total of 63 eyes from 55 keratoconus patients were randomly assigned using computer-generated randomization (www.random.org/integers) into three groups: 20 eyes in the HMW-HA group, 23 eyes in the LMW-HA group, and 20 eyes in the control group without the administration of artificial tears.

Post-CXL, the HMW-HA group received topical HMW-HA (Comfort Shield®, i.com medical GmbH, Munich, Germany) three times daily for 12 months, the LMW-HA group received topical LMW-HA (Thealose Duo®, Thea, Clermont-Ferrand, France) three times daily for 12 months, and the control group received topical polyvinyl alcohol (Refresh, Allergan, Dublin, Ireland) three times daily until epithelial defect closure. All participants underwent accelerated epithelium-off CXL (A-CXL) for 10 minutes with 9 mW/cm² ultraviolet-A irradiation. The postoperative standard treatment regimen included topical moxifloxacin (0.5% Vigamox, Alcon Inc, USA) for one week, topical dexamethasone (0.1% Dexasine-SE, Kaysersberg Pharmaceuticals, France) for one week after epithelial closure, followed by topical loteprednol 0.5% (Lotemax, Bausch & Lomb, USA) for three weeks.

Uncorrected visual acuity (UCVA), best-corrected visual acuity (BCVA), and manifest spherical equivalent (SE) were recorded at all visits. The assessment was carried out in the following order: Ocular Surface Disease Index (OSDI) questionnaire, noninvasive tear break-up time (NIBUT), corneal tomography (Pentacam, OCULUS, Wetzlar, Germany), corneal sensitivity, corneal fluorescein staining, and CCM imaging. Examinations were conducted preoperatively and at the postoperative 1th, 3rd, 6th and 12th months.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus patiens aged 18 and above who had been scheduled for corneal crosslinking

Exclusion Criteria:

* Dry eye disease, corneal thickness below 400 micrometer, pregnancy, breastfeeding, topical or systemic drug use, eye disease other than keratoconus, systemic diseases, active atopy or allergy, contact lens use, ocular surgery history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty-five patients with keratoconus were included in the study. All participants underwent accelerated epithelium-off CXL (A-CXL) for 10 minutes with 9 mW/cm² ultraviolet-A irradiation. A total of 63 eyes from 55 keratoconus patients were assigned into three groups: 17 patiens (20 eyes) in the HMW-HA group, 22 patient (23 eyes) in the LMW-HA group, and 20 patient (20 eyes) in the control group.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Corneal nerve fiber density (CNFD) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFD.
Corneal nerve fiber density (CNFD) | Postoperative 1st, 3rd, 6th and 12th months
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFD.
Corneal nerve branch density (CNBD) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNBD.
Corneal nerve branch density (CNBD) | Postoperative 1st, 3rd, 6th and 12th months
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNBD.
Corneal nerve fiber length (CNFL) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFL
Corneal nerve fiber length (CNFL) | Postoperative 1st, 3rd, 6th and 12th months
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CNFL
Corneal nerve fiber total branching density (CTBD) | Baseline
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CTBD.
Corneal nerve fiber total branching density (CTBD) | Postoperative 1st, 3rd, 6th and 12th months
  Automated tracing of nerve fibers program - CCMetrics (CCMetrics; M. A. Dabbah, ISBE, University of Manchester, Manchester, UK) was used to analyze CTBD.
Corneal Sensitivity | Baseline
  Corneal sensitivity was assessed using a Cochet-Bonnet esthesiometer (Luneau Ophtalmologue, Chartes, France).
Corneal Sensitivity | Postoperative 1st, 3rd, 6th and 12th months
  Corneal sensitivity was assessed using a Cochet-Bonnet esthesiometer (Luneau Ophtalmologue, Chartes, France).
Dendritic cell density | Baseline
  The Density of dendritic cells was calculated using ImageJ software (Image V.1.31; National Institutes of Health)
Dendritic cell density | Postoperative 1st, 3rd, 6th and 12th months
  The Density of dendritic cells was calculated using ImageJ software (Image V.1.31; National Institutes of Health)
Ocular surface disease Index (OSDI) questionnaire | Baseline
  The Turkish validated version of the OSDI, a questionnaire assesing the clinical symptoms of the ocular surface disease, was used. The 4th and 5th questions in the first section, which inquire about blurred vision and reduced vision symptoms, were excluded from the questionnaire as they could already be present in patients with keratoconus disease.
Ocular surface disease Index (OSDI) questionnaire | Postoperative 1st, 3rd, 6th and 12th months
  The Turkish validated version of the OSDI, a questionnaire assesing the clinical symptoms of the ocular surface disease, was used. The 4th and 5th questions in the first section, which inquire about blurred vision and reduced vision symptoms, were excluded from the questionnaire as they could already be present in patients with keratoconus disease.
Non invaziv tear break-up time (NI-TBUT) | Baseline
  The tear break-up time (TBUT) was evaluated non-invasively using a Sirius Scheimpflug camera (CSO, Florence, Italy).
Non invaziv tear break-up time (NI-TBUT) | Postoperative 1st, 3rd, 6th and 12th months
  The tear break-up time (TBUT) was evaluated non-invasively using a Sirius Scheimpflug camera (CSO, Florence, Italy).

SECONDARY OUTCOMES:
Visual Functions | Baseline
  Uncorrected visual acuity (UCVA), best corrected visual acuity (BCVA) by the Snellen chart, based on the logMAR scoring system and manifest spherical equivalent (SE) were assessed.
Refractive Outcomes | Postoperative 1st, 3rd and 6th months
  Uncorrected visual acuity (UCVA), best corrected visual acuity (BCVA) by the Snellen chart, based on the logMAR scoring system and manifest spherical equivalent (SE) were assessed.
Keratometric Findings | Baseline
  Corneal tomography (Pentacam, OCULUS, Wetzlar Germany) was used to obtain the data for K1, K2, Kmean, Kmax, and the Thinnest point (TP).
Keratometric Findings | Postoperative 1st, 3rd and 6th months
  Corneal tomography (Pentacam, OCULUS, Wetzlar Germany) was used to obtain the data for K1, K2, Kmean, Kmax, and the Thinnest point (TP).

CONTACTS AND LOCATIONS:
Overall Officials: Semra Akkaya Turhan, Assoc. prof., Study Chair — Marmara University
Locations (1):
- Marmara University, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozkan G, Turhan SA, Toker E. Effect of high and low molecular weight sodium hyaluronic acid eye drops on corneal recovery after crosslinking in keratoconus patients. BMJ Open Ophthalmol. 2025 Mar 29;10(1):e001890. doi: 10.1136/bmjophth-2024-001890. PMID 40157723